CLINICAL TRIAL: NCT01992159
Title: A Randomized, Double-blind, Placebo-controlled, Multi-dose Phase 2 Study to Evaluate the Efficacy, Safety and Tolerability of Romosozumab in the Treatment of Japanese Women With Postmenopausal Osteoporosis
Brief Title: Efficacy, Safety and Tolerability of Romosozumab in the Treatment of Japanese Women With Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20101291
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Postmenopausal Osteoporosis (PMO)
Keywords: Osteoporosis, Osteoporosis-Postmenopausal, Bone Diseases-Metabolic, Bone Diseases, Musculoskeletal Diseases
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Bone Diseases, Metabolic; Bone Diseases; Musculoskeletal Diseases | interventions — romosozumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo matching to romosozumab administered by subcutaneous injection once a month for 12 months.
  Interventions: Drug: Placebo
- Romosozumab 70 mg (Experimental): Participants received 70 mg romosozumab administered by subcutaneous injection once a month for 12 months.
  Interventions: Drug: Romosozumab
- Romosozumab 140 mg (Experimental): Participants received 140 mg romosozumab administered by subcutaneous injection once a month for 12 months.
  Interventions: Drug: Romosozumab
- Romosozumab 210 mg (Experimental): Participants received 210 mg romosozumab administered by subcutaneous injection once a month for 12 months.
  Interventions: Drug: Romosozumab

INTERVENTIONS:
Drug: Romosozumab — Administered by subcutaneous injection
  Other Names: AMG 785; EVENITY™
  Arms: Romosozumab 140 mg; Romosozumab 210 mg; Romosozumab 70 mg
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if treatment with romosozumab increases bone mineral density in Japanese women with postmenopausal osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

Ambulatory, postmenopausal Japanese women with osteoporosis (defined as bone mineral density T-score of ≤ -4.00 at the lumbar spine or BMD T-score of ≤ -3.50 at the total hip, or femoral neck)

Exclusion Criteria:

* Severe osteoporosis
* Use of agents affecting bone metabolism
* History of metabolic or bone disease (except osteoporosis)
* Vitamin D insufficiency (vitamin D repletion and rescreening is permitted)
* Current hyper- or hypocalcemia
* Current, uncontrolled hyper- or hypothyroidism
* Current, uncontrolled hyper- or hypoparathyroidism

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2012-10-12 (Actual); Primary Completion 2014-10-09 (Actual); Study Completion 2015-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (23):
- Japan (23):
  - Research Site, Anjyo-shi, Aichi-ken
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kitakyushu-shi, Fukuoka
  - Research Site, Yanagawa-shi, Fukuoka
  - Research Site, Mizunami-shi, Gifu
  - Research Site, Sapporo, Hokkaido
  - Research Site, Morioka, Iwate
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Saito-shi, Miyazaki
  - Research Site, Matsumoto-shi, Nagano
  - Research Site, Ueda-shi, Nagano
  - Research Site, Osaka, Osaka
  - Research Site, Takatsuki-shi, Osaka
  - Research Site, Kita-adachi-gun, Saitama
  - Research Site, Hachioji-shi, Tokyo
  - Research Site, Kiyose-shi, Tokyo
  - Research Site, Minato-ku, Tokyo
  - Research Site, Ōta-ku, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Suginami-ku, Tokyo
  - Research Site, Toshima-ku, Tokyo

REFERENCES:
- [Background] Ishibashi H, Crittenden DB, Miyauchi A, Libanati C, Maddox J, Fan M, Chen L, Grauer A. Romosozumab increases bone mineral density in postmenopausal Japanese women with osteoporosis: A phase 2 study. Bone. 2017 Oct;103:209-215. doi: 10.1016/j.bone.2017.07.005. Epub 2017 Jul 5. PMID 28687496
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 24 centers in Japan. The first participant was enrolled on 12 October 2012 and the last participant enrolled on 15 October 2013.
Pre-assignment Details: Participants were randomized in a 1:1:1:1 ratio to receive placebo or romosozumab 70, 140, or 210 mg subcutaneous (SC) injection every month (QM) for 12 months. Upon completion of the 12-month treatment period, participants were followed for another 3 months for assessment of antiromosozumab antibody formation (follow-up period).
Period: Overall Study
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Started | 63 | 63 | 63 | 63
Received Treatment | 63 | 63 | 63 | 63
Completed First 12 Months of Study | 59 | 56 | 63 | 59
Completed | 59 | 55 | 62 | 59
Not Completed | 4 | 8 | 1 | 4
Not completed — Withdrawal by Subject | 4 | 7 | 0 | 3
Not completed — Adverse Event | 0 | 1 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg | Total
Number analyzed (Participants) | 63 | 63 | 63 | 63 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (7.2) | 66.5 (6.3) | 68.4 (6.0) | 68.3 (5.9) | 67.7 (6.4)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 27 | 30 | 18 | 18 | 93
  ≥ 65 to < 75 years | 22 | 22 | 34 | 34 | 112
  ≥ 75 years | 14 | 11 | 11 | 11 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 63 | 63 | 63 | 252
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 63 | 63 | 63 | 63 | 252
Lumbar Spine Bone Mineral Density (BMD) T-score [Mean (Standard Deviation); unit: T-score] — The T-score is the bone mineral density (BMD) at the site when compared to that of a healthy thirty-year-old. Normal is a T-score of -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5; Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and a half standard deviations below the mean of a thirty-year-old man/woman.
  T-score | -2.69 (0.52) | -2.73 (0.57) | -2.65 (0.66) | -2.72 (0.42) | -2.70 (0.54)
Total Hip BMD T-score [Mean (Standard Deviation); unit: T-score] | -2.00 (0.60) | -1.97 (0.57) | -1.85 (0.68) | -1.95 (0.65) | -1.94 (0.63)
Femoral Neck BMD T-score [Mean (Standard Deviation); unit: T-score] | -2.31 (0.47) | -2.27 (0.53) | -2.28 (0.65) | -2.32 (0.59) | -2.29 (0.56)
Serum Procollagen Type 1 N-telopeptide (P1NP) [Median (Inter-Quartile Range); unit: μg/L] — Population: Participants with available data
  μg/L
    number analyzed (Participants) | 63 | 62 | 63 | 63 | 251
    (all) | 52.4 [41.9 to 62.9] | 51.9 [40.5 to 59.8] | 47.6 [37.7 to 54.9] | 50.9 [38.0 to 59.1] | 50.5 [38.6 to 59.4]
Serum Type 1 Collagen C-telopeptide (CTX) [Median (Inter-Quartile Range); unit: ng/L] | 441.0 [294.0 to 692.0] | 441.0 [289.0 to 678.0] | 374.0 [265.0 to 552.0] | 420.0 [297.0 to 690.0] | 412.0 [288.5 to 628.0]
Osteocalcin [Median (Inter-Quartile Range); unit: μg/L] | 22.17 [17.76 to 28.74] | 22.50 [17.70 to 28.46] | 21.01 [16.95 to 24.35] | 22.75 [18.07 to 27.12] | 22.03 [17.83 to 27.19]
Bone Specific Alkaline Phosphatase (BSAP) [Mean (Inter-Quartile Range); unit: μg/L] — Population: Participants with available data
  μg/L
    number analyzed (Participants) | 63 | 62 | 63 | 63 | 251
    (all) | 14.49 [12.26 to 17.56] | 13.92 [11.53 to 17.82] | 15.49 [11.85 to 17.90] | 14.72 [11.45 to 17.28] | 14.72 [11.85 to 17.75]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to 12 Months in Bone Mineral Density at the Lumbar Spine
Description: Bone mineral density was measured using dual-energy X-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging reader.
Time Frame: Baseline and 12 months
Population: Randomized participants who received at least 10 doses of the assigned randomized treatment, never received any dose of incorrect treatment, had no missing baseline values, and had at least 1 postbaseline measurement (primary efficacy subset).
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 59 | 55 | 62 | 59
percent change | 0.9 [0.1 to 1.8] | 8.4 [7.6 to 9.3] | 13.3 [12.1 to 14.5] | 16.9 [15.5 to 18.4]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 70 mg; The primary analysis was based on a repeated measures model with the percent change from baseline at months 6 and 12 in BMD of the lumbar spine as the dependent variable, and baseline BMD, machine type, interaction of baseline BMD and machine type, visit (categorical), treatment (categorical), and interaction of treatment and visit as the independent variables; using an unstructured variance covariance structure; Test type: Superiority; p < 0.0001, Repeated Measures Model — P-values were adjusted for multiplicity using a combination of a sequential test procedure and Hochberg's method to control type 1 error for the primary endpoint; Treatment Difference = 7.5, 95% CI 1-sided [lower limit 6.5]
Statistical Analysis 2: Comparison: Placebo vs Romosozumab 140 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Repeated Measures Model — [p-value comment as in outcome 1, analysis 1]; Treatment Difference = 12.4, 95% CI 1-sided [lower limit 11.1]
Statistical Analysis 3: Comparison: Placebo vs Romosozumab 210 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Repeated Measures Model — One-sided p-values were adjusted for multiplicity using a combination of a sequential test procedure and Hochberg's method to control type 1 error for the primary endpoint; Treatment Difference = 16.0, 95% CI 1-sided [lower limit 14.6]

2. Secondary Outcome: Percent Change From Baseline at 6 Months in Bone Mineral Density at the Lumbar Spine
Description: as for outcome 1
Time Frame: Baseline and 6 months
Population: Randomized participants who received at least 10 doses of the assigned randomized treatment, never received any dose of incorrect treatment, had no missing baseline values, and had at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 59 | 55 | 62 | 59
percent change | 1.2 [0.5 to 1.9] | 6.5 [5.7 to 7.2] | 10.2 [9.2 to 11.2] | 13.1 [11.7 to 14.5]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 70 mg; The analysis was based on a repeated measures model with the percent change from baseline at months 6 and 12 in BMD of the lumbar spine as the dependent variable, and baseline BMD, machine type, interaction of baseline BMD and machine type, visit (categorical), treatment (categorical), and interaction of treatment and visit as the independent variables; using an unstructured variance covariance structure; Test type: Superiority; p < 0.0001, Repeated Measures Model; Treatment Difference = 5.3, 95% CI 1-sided [lower limit 4.4]
Statistical Analysis 2: Comparison: Placebo vs Romosozumab 140 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Repeated Measures Model; Treatment Difference = 9.0, 95% CI 1-sided [lower limit 8.0]
Statistical Analysis 3: Comparison: Placebo vs Romosozumab 210 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Repeated Measures Model; Treatment Difference = 11.9, 95% CI 1-sided [lower limit 10.6]

3. Secondary Outcome: Percent Change From Baseline at 6 Months in Bone Mineral Density at the Total Hip
Description: as for outcome 1
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 59 | 55 | 62 | 59
percent change | 0.6 [-0.0 to 1.3] | 1.2 [0.5 to 2.0] | 2.3 [1.7 to 2.9] | 3.2 [2.5 to 3.9]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 70 mg; The analysis was based on a repeated measures model with the percent change from baseline at months 6 and 12 in BMD of the total hip as the dependent variable, and baseline BMD, machine type, interaction of baseline BMD and machine type, visit (categorical), treatment (categorical), and interaction of treatment and visit as the independent variables; using an unstructured variance covariance structure; Test type: Superiority; p = 0.1250, Repeated Measures Model; Treatment Difference = 0.6, 95% CI 1-sided [lower limit -0.3]
Statistical Analysis 2: Comparison: Placebo vs Romosozumab 140 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0002, Repeated Measures Model; Treatment Difference = 1.7, 95% CI 1-sided [lower limit 0.9]
Statistical Analysis 3: Comparison: Placebo vs Romosozumab 210 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Repeated Measures Model; Treatment Difference = 2.6, 95% CI 1-sided [lower limit 1.7]

4. Secondary Outcome: Percent Change From Baseline to 12 Months in Bone Mineral Density at the Total Hip
Description: Bone density was measured using dual-energy X-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging reader.
Time Frame: Baseline and 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 59 | 55 | 62 | 59
percent change | 0.6 [-0.0 to 1.3] | 2.1 [1.4 to 2.8] | 3.2 [2.6 to 3.9] | 4.7 [4.0 to 5.5]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 70 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0012, Repeated Measures Model; Treatment Difference = 1.5, 95% CI 1-sided [lower limit 0.7]
Statistical Analysis 2: Comparison: Placebo vs Romosozumab 140 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Repeated Measures Model; Treatment Difference = 2.6, 95% CI 1-sided [lower limit 1.8]
Statistical Analysis 3: Comparison: Placebo vs Romosozumab 210 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Repeated Measures Model; Treatment Difference = 4.1, 95% CI 1-sided [lower limit 3.3]

5. Secondary Outcome: Percent Change From Baseline to 6 Months in Bone Mineral Density at the Femoral Neck
Description: as for outcome 1
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 59 | 55 | 62 | 59
percent change | 0.6 [-0.1 to 1.4] | 1.0 [0.1 to 1.8] | 1.9 [1.0 to 2.9] | 3.3 [2.1 to 4.4]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 70 mg; The analysis was based on a repeated measures model with the percent change from baseline at months 6 and 12 in BMD of the femoral neck as the dependent variable, and baseline BMD, machine type, interaction of baseline BMD and machine type, visit (categorical), treatment (categorical), and interaction of treatment and visit as the independent variables; using an unstructured variance covariance structure; Test type: Superiority; p = 0.2846, Repeated Measures Model; Treatment Difference = 0.3, 95% CI 1-sided [lower limit -0.6]
Statistical Analysis 2: Comparison: Placebo vs Romosozumab 140 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0151, Repeated Measures Model; Treatment Difference = 1.3, 95% CI 1-sided [lower limit 0.3]
Statistical Analysis 3: Comparison: Placebo vs Romosozumab 210 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0001, Repeated Measures Model; Treatment Difference = 2.6, 95% CI 1-sided [lower limit 1.5]

6. Secondary Outcome: Percent Change From Baseline to 12 Months in Bone Mineral Density at the Femoral Neck
Description: as for outcome 1
Time Frame: Baseline and 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 59 | 55 | 62 | 59
percent change | 0.3 [-0.6 to 1.2] | 1.9 [1.0 to 2.7] | 2.9 [2.1 to 3.8] | 3.8 [2.7 to 4.9]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 70 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0067, Repeated Measures Model; Treatment Difference = 1.6, 95% CI 1-sided [lower limit 0.5]
Statistical Analysis 2: Comparison: Placebo vs Romosozumab 140 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Repeated Measures Model; Treatment Difference = 2.6, 95% CI 1-sided [lower limit 1.6]
Statistical Analysis 3: Comparison: Placebo vs Romosozumab 210 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Repeated Measures Model; Treatment Difference = 3.5, 95% CI 1-sided [lower limit 2.3]

7. Secondary Outcome: Percent Change From Baseline in Procollagen Type 1 N-telopeptide (P1NP)
Time Frame: Baseline, week 1, and months 1, 2, 3, 6, 9, and 12
Population: Randomized participants who received at least 10 doses of the assigned randomized treatment, never received any dose of incorrect treatment, had no missing baseline values, had at least 1 postbaseline measurement and with available data at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 59 | 55 | 62 | 59
percent change
  Week 1: number analyzed (Participants) | 59 | 54 | 62 | 59
  Week 1 | -2.5 (9.0) | 43.4 (24.0) | 65.9 (25.7) | 81.5 (34.6)
  Month 1: number analyzed (Participants) | 59 | 54 | 62 | 59
  Month 1 | -5.7 (22.1) | 32.2 (22.9) | 79.8 (41.7) | 101.6 (41.1)
  Month 2: number analyzed (Participants) | 59 | 54 | 62 | 59
  Month 2 | -10.9 (18.5) | -0.7 (18.4) | 34.6 (38.2) | 59.8 (40.5)
  Month 3: number analyzed (Participants) | 59 | 54 | 62 | 59
  Month 3 | -11.5 (20.3) | -13.1 (18.3) | 14.9 (32.2) | 25.5 (33.4)
  Month 6: number analyzed (Participants) | 59 | 54 | 62 | 58
  Month 6 | -8.9 (23.3) | -16.8 (26.0) | -2.7 (28.0) | 2.4 (24.8)
  Month 9: number analyzed (Participants) | 59 | 54 | 62 | 59
  Month 9 | -2.1 (32.0) | -16.9 (31.3) | -9.1 (30.9) | -4.0 (31.5)
  Month 12: number analyzed (Participants) | 59 | 54 | 62 | 59
  Month 12 | 4.6 (37.9) | -11.1 (29.8) | -16.2 (27.4) | -13.1 (28.1)

8. Secondary Outcome: Percent Change From Baseline in Type 1 Collagen C-telopeptide (CTX)
Time Frame: Baseline, week 1, and months 1, 2, 3, 6, 9, and 12
Population: Randomized participants who received at least 10 doses of the assigned randomized treatment, never received any dose of incorrect treatment, had no missing baseline values, had at least 1 postbaseline measurement, and with available data at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 59 | 55 | 62 | 59
percent change
  Week 1 | 11.9 (27.8) | -28.0 (25.8) | -32.1 (32.8) | -42.0 (25.4)
  Month 1: number analyzed (Participants) | 59 | 55 | 62 | 57
  Month 1 | 14.9 (40.2) | -18.0 (34.3) | -8.0 (53.9) | -24.6 (30.5)
  Month 2 | 14.1 (41.6) | -2.3 (48.4) | 14.9 (67.8) | 0.1 (49.1)
  Month 3 | 16.1 (49.0) | -5.5 (48.3) | 28.9 (84.1) | 8.1 (53.8)
  Month 6 | 13.6 (49.8) | -10.8 (52.2) | 3.2 (71.8) | -13.4 (40.6)
  Month 9 | 12.6 (56.6) | -13.2 (53.0) | -8.0 (55.7) | -15.3 (44.8)
  Month 12 | 35.4 (81.7) | -4.1 (47.2) | 2.1 (73.5) | -10.5 (53.8)

9. Secondary Outcome: Percent Change From Baseline in Osteocalcin
Time Frame: Baseline, week 1, and months 1, 2, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 59 | 55 | 62 | 59
percent change
  Week 1 | 2.6 (18.1) | 6.5 (12.6) | 7.9 (17.0) | 5.5 (14.5)
  Month 1 | -3.8 (12.7) | 26.5 (20.4) | 51.2 (31.9) | 66.4 (31.3)
  Month 2 | -7.0 (13.4) | 13.7 (15.1) | 39.3 (31.6) | 48.9 (31.6)
  Month 3 | -7.2 (16.8) | 4.9 (17.5) | 28.4 (29.7) | 27.5 (22.3)
  Month 6: number analyzed (Participants) | 58 | 55 | 62 | 58
  Month 6 | -10.3 (15.9) | -5.5 (18.8) | 10.6 (24.7) | 9.3 (19.2)
  Month 9 | -8.4 (18.2) | -6.8 (22.5) | -0.9 (24.0) | -1.3 (18.9)
  Month 12 | -6.8 (20.6) | -8.6 (21.8) | -9.4 (22.1) | -8.9 (17.9)

10. Secondary Outcome: Percent Change From Baseline in Bone Specific Alkaline Phosphatase (BSAP)
Time Frame: Baseline, week 1, and months 1, 2, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 59 | 55 | 62 | 59
percent change
  Week 1: number analyzed (Participants) | 59 | 54 | 62 | 59
  Week 1 | 1.6 (13.4) | 14.0 (14.5) | 17.0 (16.4) | 20.1 (17.9)
  Month 1: number analyzed (Participants) | 59 | 54 | 62 | 59
  Month 1 | -0.5 (22.1) | 23.0 (19.9) | 51.3 (27.6) | 66.2 (31.9)
  Month 2: number analyzed (Participants) | 58 | 54 | 62 | 59
  Month 2 | -7.8 (16.9) | 8.7 (20.8) | 31.8 (27.9) | 55.1 (31.0)
  Month 3: number analyzed (Participants) | 59 | 53 | 62 | 59
  Month 3 | -9.5 (16.3) | -2.8 (14.9) | 23.5 (26.5) | 39.6 (33.2)
  Month 6: number analyzed (Participants) | 59 | 54 | 62 | 59
  Month 6 | -6.6 (20.5) | -9.0 (19.0) | 3.1 (21.6) | 13.2 (26.8)
  Month 9: number analyzed (Participants) | 59 | 54 | 62 | 59
  Month 9 | -7.0 (20.5) | -10.7 (21.7) | -2.6 (25.3) | 3.5 (23.8)
  Month 12: number analyzed (Participants) | 59 | 54 | 62 | 59
  Month 12 | -6.3 (22.7) | -13.2 (19.9) | -13.7 (23.3) | -9.3 (21.4)

11. Secondary Outcome: Area Under the Curve Through Month 12 of P1NP
Time Frame: Baseline, week 1 and months 1, 2, 3, 6, 9, and 12.
Population: Randomized participants who received at least 10 doses of the assigned randomized treatment, had never received any dose of incorrect treatment, and had no missing P1NP measurements.
Measure: Least Squares Mean (95% Confidence Interval); unit: ug*month/L
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 59 | 54 | 62 | 58
ug*month/L | 554.5 [523.0 to 585.9] | 539.2 [506.4 to 572.0] | 638.5 [607.9 to 669.2] | 708.3 [676.6 to 740.0]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 70 mg; Test type: Superiority; p = 0.5084, ANCOVA; ANCOVA model with the AUC of P1NP at month 12 as the dependent variable, and baseline P1NP and treatment (categorical) as the independent variables; Treatment Difference = -15.3, 95% CI 2-sided [-60.8 to 30.2]
Statistical Analysis 2: Comparison: Placebo vs Romosozumab 140 mg; Test type: Superiority; p = 0.0002, ANCOVA; [statistical method as in outcome 11, analysis 1]; Treatment Difference = 84.1, 95% CI 2-sided [40.1 to 128.0]
Statistical Analysis 3: Comparison: Placebo vs Romosozumab 210 mg; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA model with the AUC of P1NP at months 12 as the dependent variable, and baseline P1NP and treatment (categorical) as the independent variables; Treatment Difference = 153.8, 95% CI 2-sided [109.2 to 198.4]

ADVERSE EVENTS:
Time Frame: 15 months
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Serious Adverse Events (participants affected / at risk) | 5/63 | 6/63 | 3/63 | 2/63
Other Adverse Events (participants affected / at risk) | 20/63 | 33/63 | 29/63 | 32/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | Romosozumab 70 mg (N=63) | Romosozumab 140 mg (N=63) | Romosozumab 210 mg (N=63)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Heat illness (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | Romosozumab 70 mg (N=63) | Romosozumab 140 mg (N=63) | Romosozumab 210 mg (N=63)
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0 | 1 | 3
Dental caries (Gastrointestinal disorders) | 1 | 4 | 3 | 2
Nasopharyngitis (Infections and infestations) | 8 | 17 | 17 | 20
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 4 | 0
Contusion (Injury, poisoning and procedural complications) | 5 | 6 | 2 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 4 | 1 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 5 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 4
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 4 | 5 | 1
Hypertension (Vascular disorders) | 2 | 1 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.